CLINICAL TRIAL: NCT05602454
Title: Virtual Care to Improve Heart Failure Outcomes (VITAL-HF) Randomized Controlled Trial
Brief Title: Virtual Care to Improve Heart Failure Outcomes (VITAL-HF)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Story Health Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00110400
Record Dates: First submitted 2022-10-27; First posted 2022-11-02 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Heart Failure With Reduced Ejection Fraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Heart Failure Medication Titration (Experimental): The Story Health platform will remotely receive daily vital signs directly from a blood pressure cuff and scale provided to the participant. Participants will also report any symptoms. All of this data will be transmitted, via the platform, to the treating clinician at the site, who will create care plans for medication titration and make clinical decisions. The care plans will be implemented with assistance from health coaches from Story Health Inc.
  Interventions: Other: Digital Heart Failure Medication Titration
- Usual Care (No Intervention): Routine clinical care will be followed. Participants will also receive a blood pressure cuff and scale, though the data will not be routinely fed back to the treating clinicians unless requested.

INTERVENTIONS:
Other: Digital Heart Failure Medication Titration — Story Health Platform, which is a remote, digital tool that provides treating clinicians collected data to make clinical decisions regarding heart failure medication titration.
  Arms: Digital Heart Failure Medication Titration

SUMMARY:
The purpose of this study is to evaluate how safe and effective a remote, digital intervention is that helps clinicians use and optimally adjust heart failure medications, compared to usual care medication use and adjustment, in participants with heart failure with reduced ejection fraction

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years of age
* Diagnosis of HF and LVEF <40% on most recent imaging assessment within 1 year prior to screening. Any validated method for assessing LVEF may be used for enrollment including echocardiogram, cardiac magnetic resonance imaging, etc. For participants with an LVEF reported qualitatively (e.g., moderate LV dysfunction) or as a range on the most recent imaging assessment that includes 40% (e.g., 35-45%), then the site investigator should review the imaging study and determine if the participant has an LVEF <40%. Participants with a new diagnosis of HFrEF may be enrolled. The enrollment will be monitored to ensure no more than 50% of the total cohort have new-onset HFrEF.
* Access to a smartphone including through a family member of caregiver
* Fluent in written and spoken English

Exclusion Criteria:

* Optimized or nearly-optimized on evidence-based medical therapies for HFrEF as determined by local investigator.
* Current pregnancy
* Chronic use of intravenous inotropic medications including milrinone, dobutamine, or dopamine
* eGFR of <20 mL/min/1.73m2 or ongoing chronic dialysis at screening
* Prior heart transplant
* Current or planned left ventricular assist device
* Currently receiving hospice care
* Chronically resides in an assisted living or skilled nursing facility where food and medications are managed by facility personnel
* Terminal illness other than HF with a life expectancy of less than 1 year as determined by the enrolling clinician-investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2022-12-02 (Actual); Primary Completion 2025-03-05 (Actual); Study Completion 2025-03-05 (Actual)

PRIMARY OUTCOMES:
Change in medical therapy, as measured by the Heart Failure Medical Therapy Score | Baseline, 6 months
  Scores are 0-3 for 7 key medication classes for heart failure with reduced ejection fraction where 0 represents no use of the medication class

SECONDARY OUTCOMES:
Change in medical therapy, as measured by the Kansas City Medical Optimization score | Baseline, 6 months
  Scores are the average of the total daily dose to target dose values for HF medications. Scores range from 0-100.
Intensification of evidence-based medical therapies, measured by number of participants with reported changes. | baseline, 6 months
  Proportion of participants with any intensification of and cumulative number of intensifications of evidence-based medical therapies for HFrEF from baseline to last follow-up.
Proportion of participants on 50% of published target doses of evidence-based medical therapies for HFrEF at last follow-up. | 6 months
  The last measure dose will be compared with the target dose in the 2022 Heart Failure Guidelines.
Proportion of participants on 100% of published target doses of evidence-based medical therapies for HFrEF at last follow-up. | 6 months
  The last measure dose will be compared with the target dose in the 2022 Heart Failure Guidelines.
Combined Emergency department visits and hospitalizations, as measured by number of subjects with at least one occurrence | 3 months, 6 months
  Combined Emergency department visits and hospitalizations related to evidence-based medical therapies for HFrEF including symptomatic hypotension, hyperkalemia, and angioedema

OTHER OUTCOMES:
Change in participant-reported medication adherence using the Voils score | Baseline, 6 months
  The Voils score includes questions used to assess medication adherence. Answers range between "not at all" and "very much", with 3 options in between. "Not at all" means a dose was not missed and "Very much" means dose was missed for that reason.
Change in Kansas City Cardiomyopathy Questionnaire Overall Summary score | Baseline, 6 months
  The Kansas City Cardiomyopathy Questionnaire 12-item version includes multiple domains: symptom frequency, quality of life, social limitation, and physical limitation. The Overall Summary score incorporates the averages of these 4 domains and is reported on a 0-to-100-point scale, where lower scores represent more severe symptoms and/or limitations and scores of 100 indicate no symptoms, no limitations, and excellent quality of life.
Global rank score across 3 hierarchical tiers of a composite outcome: time to death, time to HF hospitalization, change from baseline to last follow-up in the HF medical therapy score | baseline, 6 months
Composite of all-cause death and total worsening HF events defined by hospitalizations for acute HF and urgent HF events | 3 months, 6 months
Worsening HF events defined by hospitalizations for acute HF and urgent HF events | 3 months, 6 months
All-cause hospitalizations | 3 months, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Adam DeVore, MD, Principal Investigator — Duke University
Locations (7):
- United States (7):
  - Cardiovascular Institute of Northwest Florida, Panama City, Florida
  - Ascension St. Vincent, Indianapolis, Indiana
  - The University of Kansas Medical Center, Kansas City, Kansas
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Saint Luke's Health Systems, Kansas City, Missouri
  - Duke University, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khan MS, Sauer AJ, Green CL, McDermott J, Khan MS, Chaudhry SP, Haghighat AR, Bennett MK, Martyn T, Shah H, Govil A, Stanis T, Albert NM, DeVore AD. Rationale, design, and baseline characteristics of the virtual care to improve heart failure outcomes (VITAL-HF) trial. Am Heart J. 2025 Dec;290:46-57. doi: 10.1016/j.ahj.2025.06.001. Epub 2025 Jun 3. PMID 40473009